CLINICAL TRIAL: NCT04214600
Title: Brief Cognitive Behavioral Therapy for Adherence and Depression in Patients With Type 2 Diabetes in an Urban Primary Care Facility: Randomized Controlled Trial
Brief Title: Cognitive Behavioral Therapy for Adherence in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadine Mansour, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBT for T2D
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes; Depression
Keywords: Type 2 diabetes; Depression; Treatment adherence; Cognitive behavioral therapy; Randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Treatment Adherence and Compliance | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, parallel-group, two-arm controlled trial
Who Masked: Participant
Masking Description: Blinding of patients and all members of the research team (except for the researcher conducting the CBT intervention) will be carried out throughout the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): This group will receive four CBT sessions twice a month for two months
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Control (No Intervention): This group will be scheduled the same number of visits as a follow up for diabetes

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Patients in the CBT intervention group will receive four educational sessions for 30-45 minutes on one to one basis every two weeks during patients' regular follow up visits. The visits will be scheduled depending on the patient's availability. The sessions will be delivered by a trained physician. The sessions will include:
  Session 1: Dealing with thoughts of sadness and depression Session 2: Dealing with thoughts of anxiety and stress Session 3: Dealing with anger Session 4: Enhancement of coping and problem-solving skills
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Despite the significant relationship between depression and diabetes, there are few published studies testing the effect of cognitive behavioral therapy in improving disease outcomes among diabetics in primary healthcare settings in Egypt. The study aims at assessing the efficacy of cognitive behavioral therapy combined with diabetes education versus control receiving diabetes education alone in helping patients with Type 2 Diabetes and depressive symptoms to achieve glycemic control and compliance to treatment.

DETAILED DESCRIPTION:
The psychological status of diabetic patients impacts their health behavior and clinical outcomes significantly. Psychological interventions are important tools to amending health behavior in Type 2 Diabetes (T2D). Cognitive Behavioral Therapy (CBT) has been an effective non-pharmacologic treatment for a wide variety of mental disorders such as depression, anxiety, post-traumatic stress disorder, eating disorders, and schizophrenia. The therapeutic approach promotes coping capabilities against difficult situations. It targets a change in negative patterns of cognition and associated behaviors and promotes emotional regulation.

Depression in diabetic patients is under-recognized. It is estimated that 44% of depressed patients are recognized by practitioners. Such lack of recognition is attributed to poor diabetic outcomes. There is a growing body of research that explores the effectiveness of this psychological technique in managing chronic physical diseases. Despite the success of CBT in managing psychiatric morbidities, research on its use in the treatment of diabetes is limited and with varying results. Moreover, the majority of studies that have investigated the burden of depression in T2D have been carried out in high-income countries, but little is done in the Middle East and North Africa (MENA) region especially Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the American Diabetes Association (ADA) criteria for T2D (glycated hemoglobin (HbA1c) ≥6.5%, fasting glucose ≥126mg/dL) with diagnosis confirmed by the participants' medical clinicians.
* Participants aged more than 35 years; ambulatory; able to give informed consent; and able to obtain reliable information.
* Eligible patients will be screened for depressive symptoms using the Beck Depression Inventory (BDI). They will be included if they score 11-30 based on BDI (Mild mood disturbance to Moderate depression).

Exclusion Criteria:

* Participants will be excluded if they have type I diabetes and psychiatric disorders other than mood or personality disorders. Depressed patients on treatment for depression will not be included.
* Suicidal patients and those diagnosed with major depressive disorder will be referred to a psychiatrist.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Mansour, MD, Principal Investigator — Al-Agouza Family Medicine Center & Faculty of Medicine, Cairo University
Locations (1):
- Al-Agouza Family Medicine Center (AFMC)., Agouza, Giza Governorate, Egypt

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Therapy: This group will receive four CBT sessions twice a month for two months
  Cognitive Behavioral Therapy (CBT): Patients in the CBT intervention group will receive four educational sessions for 30-45 minutes on one to one basis every two weeks during patients' regular follow up visits. The visits will be scheduled depending on the patient's availability. The sessions will be delivered by a trained physician. The sessions will include:
  Session 1: Dealing with thoughts of sadness and depression Session 2: Dealing with thoughts of anxiety and stress Session 3: Dealing with anger Session 4: Enhancement of coping and problem-solving skills
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy | Control
Started | 50 | 50
Completed | 41 | 36
Not Completed | 9 | 14
Not completed — Lost to Follow-up | 9 | 14

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Behavioral Therapy: This group will receive four CBT sessions twice a month for two months
  Cognitive Behavioral Therapy (CBT): Patients in the CBT intervention group will receive four educational sessions for 30-45 minutes on one to one basis every two weeks during patients' regular follow up visits. The visits will be scheduled depending on the patient's availability. The sessions will be delivered by a trained physician and will include:
  Session 1: Dealing with thoughts of sadness and depression Session 2: Dealing with thoughts of anxiety and stress Session 3: Dealing with anger Session 4: Enhancement of coping and problem-solving skills
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Count of Participants; unit: Participants]
  Age interval: 35-44 | 5 | 12 | 17
  Age interval: 45-54 | 19 | 18 | 37
  Age interval: 45-64 | 11 | 6 | 17
  Age interval: ≥65 | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 34 | 35 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change of Glycated Hemoglobin A1c (Hb A1c) After the Cognitive Behavioral Therapy Sessions
Description: Assess the effect of the CBT combined with diabetes education versus control receiving diabetes education alone on glycemic measures of patients with T2D and depression
Time Frame: Baseline and 3 months
Population: Of the 100 patients that met the inclusion criteria and completed the baseline assessment, only 77 patients completed the post-intervention assessment.
Measure: Mean (Standard Error); unit: percent
Groups:
- CBT Group: Participants received four Cognitive Behavioral Therapy sessions and diabetes education
- Control Group: Participants received diabetes education only
Arm/Group | CBT Group | Control Group
Number analyzed (Participants) | 41 | 36
percent | 7.70 (0.23) | 8.42 (0.25)

2. Secondary Outcome: Change of Depression Score on Beck's Depression Index
Description: Assess the effect of the CBT combined with diabetes education versus control receiving diabetes education alone on depressive symptoms of patients with T2D and depression
  (Beck's Depression Index scores range between 1-40 where high scores mean worsening outcome and low scores mean improving outcome)
Time Frame: baseline and 3 months
Population: Of the 100 patients that met the inclusion criteria and completed the baseline assessment, only 77 patients completed the post intervention assessment.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Control Group: Participants received four diabetes education only
Arm/Group | CBT Group | Control Group
Number analyzed (Participants) | 41 | 36
score on a scale | 12.25 (1.09) | 16.49 (1.16)

ADVERSE EVENTS:
Time Frame: 6 months (time is calculated from the first CBT session/appointment up to 3 months post-intervention).
Groups:
- CBT Group: Participants received four CBT sessions and diabetes education
Arm/Group | CBT Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Shortage of HbA1c preparation kits. Retention of participants was a challenge although visits were scheduled at patients' convenience.

The study was conducted in one healthcare center. Long term effect of the intervention was not examined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT04214600/Prot_SAP_000.pdf